CLINICAL TRIAL: NCT01674972
Title: Glucose-induced Glucagon-like Peptide 1 (GLP-1) Secretion in NAFLD Patients Compared to Healthy Controls
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: EKBB 224/02.2
Record Dates: First submitted 2012-08-24; First posted 2012-08-29 (Estimated); Last update posted 2012-08-29 (Estimated); Status verified 2012-08

CONDITIONS: Non Alcoholic Fatty Liver Disease; Non Alcoholic Steatohepatitis
Keywords: NAFLD; NASH; GLP-1
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Glucose Tolerance Test

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- NAFLD: Patients with biopsy proven NAFLD
  Interventions: Other: Oral glucose tolerance test
- Control: Matched healthy control subjects
  Interventions: Other: Oral glucose tolerance test

INTERVENTIONS:
Other: Oral glucose tolerance test — Oral intake of 75 g glucose after overnight fast

SUMMARY:
The incretin effect is impaired in patients with type 2 diabetes mellitus (T2DM), thus GLP-1 receptor agonists are used for the treatment of T2DM. Insulin resistance is a pathophysiologic hallmark of non-alcoholic fatty liver disease (NAFLD). The incretin effect in patients with NAFLD has not been studied. The aim of this study is to quantify GLP-1 secretion in response to oral glucose tolerance test (oGTT) in patients with NAFLD compared to healthy controls. The results of this study will expand the knowledge of the pathophysiology of NAFLD and serve as a rational for potential future treatment strategies.

DETAILED DESCRIPTION:
Primary endpoint: GLP-1 response to oral glucose Secondary endpoints: glucose and insulin responses to oral glucose challenge

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven NAFLD or NASH

Exclusion Criteria:

* additional concomitants liver disease
* T2DM
* alcohol consumption >40g/d for male subjects and >20g/d for female subjects

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with biopsy proven NAFLD and NASH will be recruited from the Hepatology Outpatient Clinic, Division of Gastroenterology and Hepatology, University Hospital Basel.
  Healthy control subjects will be matched to NAFLD and NASH patients.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2011-01; Primary Completion 2012-04 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Glucagon-like Peptide 1 (GLP-1) secretion in response to oGTT | 0, 15, 30, 60, 90, 120 min. after glucose administration
  The difference in GLP-1 secretion in response to oGTT as assessed by area under the curve (AUC) and peak plasma concentration (cmax) in patients with NAFLD compared to healthy controls.

SECONDARY OUTCOMES:
Insulin secretion and glucose curves in response to oGTT | 0, 15, 30, 60, 90, 120 min. after glucose administration

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Beglinger, MD, Principal Investigator — University Hospital Basel, Division of Gastroenterology and Hepatology
Locations (1):
- University Hospital Basel, Division of Gastroenterology and Hepatology, Basel, Switzerland